CLINICAL TRIAL: NCT06894836
Title: Hybrid Type 2 Implementation-Effectiveness Trial of a Third Wave Virtual Reality Treatment for Youth Depression and Anxiety
Brief Title: Hybrid Type 2 Implementation-Effectiveness Trial of a Third Wave Virtual Reality Treatment for Youth Depression/Anxiety
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Orygen (Other)
Responsible Party: Principal Investigator, Imogen Bell, Senior Research Fellow & Psychologist, Principal Investigator, PhD (Clin Psych), Orygen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31083; BFG012 (Other Grant/Funding Number: Queensland Mental Health Commission Better Futures grant)
Record Dates: First submitted 2025-03-14; First posted 2025-03-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Depression Anxiety Disorder
Keywords: Virtual reality; Acceptance and commitment therapy; Youth mental health; Depression; Anxiety; Psychological intervention
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single arm hybrid type 2 implementation-effectiveness trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Third wave VR intervention
  Interventions: Behavioral: Third wave VR therapy

INTERVENTIONS:
Behavioral: Third wave VR therapy — All participants in this trial will receive the VR intervention which is adapted from third wave CBT protocols (including mindfulness and Acceptance and Commitment Therapy) and focuses on decentering-the ability to step back and view thoughts and emotions as temporary, objective events rather than identifying with them. Decentering has been linked to improved emotional regulation, reduced rumination, and better psychological flexibility, which in turn can lead to improvements in depression and anxiety symptoms. The intervention is clinician-delivered in a clinical setting, one-on-one, over 4-5 sessions (60 min each) across 10-12 weeks. Each session includes psychoeducation, a 15-minute VR experience, and debriefing. Sessions cover three core techniques targeting improvement in decentering ability: 1) arousal reduction via controlled breathing, 2) sitting with discomfort without reacting, and 3) cognitive defusion by changing perception of negative thoughts.

SUMMARY:
This research will evaluate a new virtual reality (VR) intervention to support youth with depression and anxiety. While VR has shown promise for adult mental health, little is known about its use in youth or routine clinical care. The VR intervention is based on Acceptance and Commitment Therapy (ACT) and immerses young people in fun, engaging environments to teach practical coping skills for managing distress. Clinicians within youth mental health services will use the VR intervention within their routine treatment of young people. The study will evaluate both the preliminary effectiveness of the VR intervention for improving youth mental health, as well as real-world implementation outcomes to understand how it can be successfully adopted in clinical settings. The trial will use a single-group, pre-post design, with treating clinicians delivering the intervention to up to 75 young people seeking treatment for depression and anxiety over a 12-week period. Assessments will be conducted at baseline, immediately after the intervention (12 weeks), and four weeks post-intervention (16 weeks).

DETAILED DESCRIPTION:
Youth mental ill-health is a global crisis. One in five young people experience a mental health disorder every year, and suicide is a leading cause of death in this age group. In addition to costing the global economy $1 trillion per year in lost productivity, mental ill-health can have a severe and long-lasting impact on the lives of young people. Despite this, only a small proportion receive access to care, and of those that do, most fail to fully recover.

Technology has the potential to overcome many systemic barriers to accessing quality, sustainable care and importantly provide treatments tailored to young people's needs. In particular, virtual reality (VR) treatments have potential to tackle key limitations in youth mental health care. Through a VR headset, young people are transported into virtual environments that can provide powerful therapeutic experiences, enabling them to learn and practice skills to overcome mental health symptoms within personally relevant situations, under the safe and controlled supervision of a clinician. As a highly novel and interactive digital medium, VR has capacity to address barriers to help seeking and poor engagement amongst young people by delivering treatments that are fun, interesting and memorable. Meta analyses of randomised controlled trials have clearly supported the efficacy of VR treatments for improving mental health outcomes, however there are currently no available evidence-based options for youth and no studies have examined how VR treatments can be implemented in real world settings. This is a clear gap, with research demonstrating there is interest and need amongst clinicians and young people for innovative digital tools like VR to improve clinical care.

Through co-design with young people with lived experience and clinicians, a new VR treatment has been developed for youth depression and anxiety. Depression and anxiety are core transdiagnostic symptoms prominent in mood and anxiety disorders, which represent the most prevalent and debilitating mental health conditions with the highest burden of disease in youth populations. This new VR treatment is a blended clinical support tool which harnesses immersive VR environments to deliver targeted evidence-based treatment for depression and anxiety. Through engaging, interactive exercises, young people are guided to learn and practice core psychological skills based on ACT, an evidence-based treatment for youth depression and anxiety. Clinicians can use the third wave VR intervention within therapy sessions to help young people learn and practice these core skills in an engaging way, providing opportunities to improve treatment engagement, reduce drop out, and deliver a more effective learning experience that can translate into greater improvements in depression and anxiety in the real world.

Previous studies by our group included interviews with 30 young people and 10 clinicians which highlighted the perceived value of the third wave VR treatment for supporting clinical treatment by improving engagement and supporting therapeutic learning. An early experimental study [under review] with 20 young people found that a single session of MIND could improve negative mood states, with 100% of the sample preferring it to traditional therapy methods. As a next phase in this research, the current project aims to conduct a hybrid type 2 effectiveness-implementation trial to establish proof-of-concept evidence that the MIND intervention can be used to treat youth depression and anxiety within a routine youth mental health service setting. This trial design enables the simultaneous testing of implementation and effectiveness outcomes, thus accelerating the research to translation pipeline by seeking to understand how interventions can be implemented in real world settings.

The aims of this single-arm hybrid effectiveness-implementation pilot study are to:

1. Assess the feasibility of the study protocol, including recruitment, retention, trial-related adverse events, and assessment completion.
2. Evaluate the feasibility and acceptability of implementing the MIND intervention within routine youth mental health care settings, with a focus on intervention delivery, fidelity to the intervention model, and satisfaction levels among both participants and clinicians.
3. Identify barriers and facilitators to implementing the MIND intervention in routine care settings, including implementation indicators relating to staff training, resource availability for delivery, organisational support, clinician perceptions, and logistical barriers and facilitators.
4. Explore the preliminary effectiveness and safety of the MIND intervention by assessing changes over time in clinical outcomes, including measures of depression, anxiety, intervention mechanisms, quality of life, and intervention-related adverse events.

ELIGIBILITY:
There are three populations recruited for this trial:

INCLUSION CRITERIA

Young people

1. Aged between 12-25 years (inclusive)
2. Current client of a participating youth mental health service
3. Seeking or receiving treatment for depression and/or anxiety
4. Sufficient command of the English language

Clinicians Employed at a participating youth mental health service and involved in the delivery of psychological treatment of young people presenting with depression and anxiety

Service staff Work within a participating youth mental health service in a leadership (team lead or service manager) or administrative role.

EXCLUSION CRITERIA:

Young people

1. Moderate or severe audio or visual condition precluding engagement with the VR equipment (assessed on a case-by-case basis)
2. Counter indication based on clinical judgement e.g., active suicidal risk or intellectual disability.

Clinicians Unable to commit to delivering the MIND intervention (5 sessions over 10-12 weeks).

Service staff Nil

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility - recruitment and retention rates | Baseline
  Rates of how many participants sign up and are enrolled in the program, along with the drop-out rate throughout the program.
Acceptability - intervention endorsement | 12 weeks post intervention commencement
  Proportion of respondents who state they would recommend the intervention to other young people, measured using a purpose built self-report acceptability questionnaire. 1-5 scale, higher scores indicate higher likelihood or recommending to others.
Effectiveness - severity of depression | Baseline, 12 weeks post intervention commencement, 16 week post intervention commencement (follow up)
  Mean pre-post scores, effect sizes and associated confidence intervals for the severity of depression assessed by the Patient Health Questionnaire-8 (PHQ-8). Range 0-28, higher indicates more severe depression.
Effectiveness - severity of anxiety | Time Frame: Baseline, 12 weeks post intervention commencement, 16 week post intervention commencement (follow up)
  Description: Mean pre-post scores, effect sizes and associated confidence intervals for the severity of anxiety assessed by the Generalized Anxiety Disorder-7 (GAD-7). Range 0-28, higher indicates more severe anxiety.

SECONDARY OUTCOMES:
Adverse events | Baseline, 12 weeks post intervention commencement, 16 week post intervention commencement (followup)
  The number of serious adverse events specifically related to the intervention or trial
Feasibility - attendance rates of assessments and sessions | 12 weeks post intervention commencement
  Record of attendance via audit of attendance logs
Feasibility - VR utilisation | 12 weeks post intervention commencement
  Number and proportion of sessions within the intervention period in which VR was used within intervention sessions.
Feasibility - intervention implementation | 12 weeks post intervention commencement
  Feasibility of Implementation Measure [FIM] (completed by service staff and clinicians)
Acceptability - intervention satisfaction | 12 weeks post intervention commencement
  Theoretical Framework of Acceptability Questionnaire (TFAQ) completed by young people, clinicians and service staff. Range 19-95, higher scores indicate greater acceptability.
Acceptability - therapeutic alliance | 12 weeks post intervention commencement
  Working Alliance Inventory-Short Revised (WAI-SR). Range 12-60, higher scores indicating better working alliance between therapist and client.
Acceptability - cybersickness within headset | Within each intervention session
  Average score on single item captured within VR headset during sessions requiring respondents toindicate the extent to which they felt uncomfortable, sick or dizzy (0 not at all to 10 very much)
Acceptability - VR presence | Within each intervention session
  Average score on single item captured within VR headset during sessions requiring respondents to indicate the extent to which they felt present in the VR environment (0 not at all to 10 very much)
Implementation - adoption | 12 weeks post intervention commencement
  Proportion of trained clinicians who implement MIND during the trial period.
Implementation - fidelity | Measured during monthly meetings with services, during training sessions (immediately following clinician recruitment), monthly supervision sessions, and each time a support ticket is logged
  Number of and attendance at, 1) facilitation meetings with services, 2) training sessions, and 3) supervision sessions, as well as number of technical support calls.
Effectiveness - emotional distress | Baseline, 12 weeks post intervention commencement, 16 week post intervention commencement (follow up)
  Kessler Psychological Distress Scale (K10). Range 10-50, higher indicates more severe emotional distress.
Effectiveness - severity of repetitive negative thinking | Baseline, 12 weeks post intervention commencement, 16 week post intervention commencement (followup)
  Perseverative Thinking Questionnaire (PTQ). Range 0-60, higher indicates more severe repetitive negative thinking.
Effectiveness - trait decentering | Baseline, 12 weeks post intervention commencement, 16 week post intervention commencement (followup)
  Metacognitive Processes of Decentering-Trait (MPoD-t). Range 15-75, higher scores indicate greater decentering ability.
Effectiveness - state decentering | Measured within VR headset before and after each therapeutic exercise
  Metacognitive Processes of Decentering-State (MPoD-s). Range 0-30, higher score indicates greater decentering in the moment.
Effectiveness - cognitive defusion | Baseline, 12 weeks post intervention commencement, 16 week post intervention commencement (followup)
  Cognitive Fusion Questionnaire (CFQ)
Effectiveness - psychological inflexibility | Baseline, 12 weeks post intervention commencement, 16 week post intervention commencement (followup)
  Avoidance and Fusion Questionnaire - Youth (AFQ-Y). Range 0-32, higher scores indicate greater psychological inflexibility.
Effectiveness - quality of life | Baseline, 12 weeks post intervention commencement, 16 week post intervention commencement (followup)
  Assessment of Quality-of-Life Scale (AQoL-6D) Adolescent. Score range from 0-1, higher scores indicate better quality of life.
Effectiveness - wellbeing | Baseline, 12 weeks post intervention commencement, 16 week post intervention commencement (followup)
  Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). Range 14-70, higher scores indicating better wellbeing.
Implementation - number and types of implementation determinants | Measured during monthly supervision meetings, all scheduled and unscheduled meetings, when a support ticket is logged, and end of study interviews with service staff, clinicians and young people (up to 1 year)
  Captured through process data related to clinical supervision and other study engagement points with participating clinicians and service staff (i.e. de-identified notes from supervision sessions, technical assistance calls, and research meetings), and via qualitative interviews with service staff , clinicians, and young people at the end of their involvement with the study.
Implementation - clinician confidence and competence | Immediately pre and post training, which occurs within 2 weeks of recruitment and consent of clinicians at the start of the study
  Purpose-built scale (no title or acronym) capturing self-rated confidence and competence by clinicians. Scale items range 1-4, higher indicating stronger confidence and competence.

CONTACTS AND LOCATIONS:
Overall Officials: iMOGEN H Bell, PhD, Principal Investigator — Orygen

IPD SHARING:
Plan to Share IPD: No
Those interested in accessing data can contact the researchers directly to discuss this.